CLINICAL TRIAL: NCT05218161
Title: Comparing the Hemodynamic Effect of Dexmedetomidine Alone With Dexmedetomidine Plus Ketamine Combination in Post Cardiac Surgery Patients: A Randomized Controlled Trial
Brief Title: Hemodynamic Effect of Dexmedetomidine Alone With Dexmedetomidine Plus Ketamine Combination in CABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chaudhry Pervaiz Elahi Institute of Cardiology (Other Government)
Responsible Party: Principal Investigator, Shumaila rai, Consultant anesthetist, Chaudhry Pervaiz Elahi Institute of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CPEIC No. 153; 153 (Registry Identifier: CPEIC)
Record Dates: First submitted 2022-01-18; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Hemodynamic Instability
Keywords: Cardiac Surgery; Dexmedetomidine; Extubation; Hemodynamics; Ketamine; Fentanyl
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DA (Active Comparator): Group DA: will be assigned to patients in whom dexmedetomidine alone will be used.
  Interventions: Drug: Dexmedetomidine alone
- KD (Experimental): Group KD: will be assigned to patients receiving ketamine plus dexmedetomidine.
  Interventions: Drug: Dexmedetomidine alone

INTERVENTIONS:
Drug: Dexmedetomidine alone — All the patients in group DA will be sedated using dexmedetomidine 1mcg/kg IV bolus, followed by 0.3-0.7mcg/kg/h infusion to maintain Ramsay sedation score ≥4 during assisted ventilation.

SUMMARY:
In post cardiac surgery, many cardiovascular and other complications may occur that lead to increase in mortality and hospital stays. Meticulous perioperative management is important to avoid these adverse events. Tachycardia is the main cause of post coronary artery bypass graft (CABG) myocardial ischemia which can be decreased by sedation and analgesia.

DETAILED DESCRIPTION:
Dexmedetomidine is a highly specific alpha 2 adrenoreceptor agonist. Its sedative effect results from stimulation of alpha 2 adrenoreceptors in the central nervous system (in the locus coeruleus) independent of GABA system contrary to other drugs.Dexmedetomidine has better sedative effect and similar respiratory and hemodynamic effects to midazolam. It does not depress respiratory drive or decrease arterial oxygen saturation so intravenous (IV) continuous sedation with dexmedetomidine does not change the normal course of ventilator weaning and extubation. It produces a unique EEG pattern of sleep that closely resembles that of normal physiological sleep that allows easy arousal. Dexmedetomidine also has analgesic effect. All these properties make dexmedetomidine a first line drug for the cooperative sedation management in the Intensive Care Unit (ICU). Ketamine is a phencyclidine nonbarbiturate derivative that binds with N methyl d aspartate and sigma opioid receptors to produce dissociative anesthesia, analgesia, and amnesia with little or no respiratory or cardiovascular depression. Ketamine inhibits endothelial nitric oxide production leading to positive inotropic action and vasoconstriction which preserves hemodynamic stability. Dexmedetomidine can effectively and safely attenuate the ketamine induced hemodynamic pressor response and psychomimetic effects. Dexmedetomidine expected to prevent the tachycardia, hypertension, salivation, and emergence phenomena associated with ketamine. Ketamine may prevent the bradycardia and hypotension that have been reported with dexmedetomidine. Review of literature has shown that there are very few studies present on the comparison of combination of Ketamine and dexmedetomidine with dexmedetomidine alone especially in post cardiac surgery patients and therefore further studies are required to ascertain the role of dexmedetomidine in terms of hemodynamic effects after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients of 40-60 years old Hemodynamically stable with normal or moderately impaired left ventricular function Ejection fraction >40% that underwent elective surgery CABG surgery for single vessel

Exclusion Criteria:

Hemodynamic instability intraoperative. Patients on moderate to high vasopressors or ionotropes. Ejection fraction less than 40%. Off pump surgery. Patient on mechanical supports.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic stability | 06 months
  Hemodynamic stability:If blood pressure and heart rate are with in appropriate limits,it will be considered as hemodynamically stable.
  Blood pressure:MAP>65 mmhg is considered stable. Heart rate:80-100 bpm is considered stable.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shumaila Rai, FCPS, Principal Investigator — Chaudhry Pervaiz Elahi Institute of Cardiology
Locations (1):
- CPEIC, Multan, Pakistan

IPD SHARING:
Plan to Share IPD: No